CLINICAL TRIAL: NCT06292858
Title: A Phase Ia Study to Evaluate the Safety/Tolerability, Pharmacokinetics and Preliminary Efficacy of IMB071703 Injection in Patients With Recurrent or Metastatic, Advanced Solid Tumors
Brief Title: Safety/Tolerability, PK and Efficacy of IMB071703 Injection in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijng Immunoah Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMB071703-101
Record Dates: First submitted 2024-02-20; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Recurrent or Metastatic, Advanced Solid Tumors
MeSH Terms: conditions — Recurrence; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Part A: Dose escalation phase
  Six dose levels of IMB071703 injection are planned in Part A, 1 subject in the first dose level (accelerated titration design), 3 subjects in the 2nd through 6th dose levels separately (conventional Fibonacci 3+3 design). 19 to 33 subjects are expected to enroll.
  Part B: Dose/cohort expansion phase
  1 to 2 dose levels of subjects with 1 to 2 tumor types are tentatively planned; a total of up to 15 subjects are included in each dose level for each tumor type, 15 to 60 subjects are expected to enroll.
  Interventions: Drug: IMB071703 injection

INTERVENTIONS:
Drug: IMB071703 injection — Intratumoral injection

SUMMARY:
A Phase Ia Study to Evaluate the Safety/Tolerability, Pharmacokinetics and Preliminary Efficacy of IMB071703 Injection in Subjects with Recurrent or Metastatic，Advanced Solid Tumors

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participating in this clinical study and signing a written informed consent form and being able to comply with clinical visits and study-related procedures.
2. Male or female subjects ≥ 18 and ≤ 75-year age when signing the informed consent form.
3. Expected survival time of not less than 3 months (as judged by the investigator)
4. Subjects with histologically or cytologically confirmed advanced malignant solid tumors, ie, recurrent or metastatic, advanced solid tumors, who have failed the standard therapy or who are not suitable for standard therapy at this stage.
5. Subjects are able to provide tumor tissue samples (archived tumor tissue within one year as much as possible or fresh specimens of core needle aspiration).
6. According to RECIST V1.1 criteria, (dose escalation phase), at least one evaluable tumor lesion; (dose expansion phase) at least one measurable tumor lesion (tumor lesions located in the previously radiotherapy area or other localized regional treatment area are generally not considered measurable unless the lesion has clearly progressed or persists after three months of radiotherapy).
7. Patients are required to have injectable lesions that meet the current dosage administered in the dose level. Superficial lesions are preferred, and deep lesions that can be injected under the ultrasound/CT guidance [injectable lesions cannot have previously been treated with radiotherapy or other intratumoral injections, and lesions with a high risk of bleeding (eg, adjacent to large blood vessels, the presence of large blood vessels in the tumor or vascular encasement) should not be considered injectable lesions].
8. Eastern Cooperative Oncology Group (ECOG) physical performance score 0-1.
9. Bone marrow reserve and organ function must meet the following requirements (no blood transfusion and no supportive treatment with blood components or granulocyte colony cytokines within 14 days before the first treatment).

Exclusion Criteria:

Subjects with any of the following conditions are not eligible for this study:

1. Received or are receiving any anti-CD40 and/or CD137 therapy.
2. Subjects who have received or plan to receive allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation/bone marrow transplantation.
3. Patients with active autoimmune diseases
4. Used live attenuated vaccines within 4 weeks before the first dosage of study drug.
5. Received immunotherapy and experienced ≥ Grade 3 irAEs or ≥ Grade 2 immune-related myocarditis.
6. Used immunomodulatory drugs within 14 days before the first dosage of study drug, including but not limited to thymosin, interleukin-2, interferon, etc.
7. Received systemic corticosteroids (prednisone > 10 mg/day or equivalent dosage of similar drug) or other immunosuppressive agents within 14 days before the first dosage of study drug (except for the following: topical, ocular, intra-articular, intranasal, and inhaled corticosteroids are allowed; short-term use of corticosteroids for prophylaxis, eg, to prevent contrast agent from allergy).
8. Received anti-tumor therapy such as systemic chemotherapy, radiotherapy, targeted therapy, endocrine therapy, biological therapy and immunotherapy within 4 weeks before the first dosage of study drug, except for the following items: nitrosourea or mitomycin C within 6 weeks before the first dosage of study drug; oral fluoropyrimidines, small-molecule targeted drugs and traditional Chinese medicines with anti-tumor indications within 2 weeks before the first dosage of study drug; local palliative radiotherapy within 2 weeks before the first dosage of study drug;
9. Received other unmarketed study drugs or treatments within 4 weeks before the first dosage of investigational drug.
10. Received major organ surgery (excluding diagnostic needle biopsy treatment) or significant trauma within 4 weeks before the first dosage of study drug, or the need for elective surgery during the study.
11. Serious wounds/ulcers/fractures that cannot be healed within 4 weeks before the first dosage of study drug.
12. The adverse events caused by previous anti-tumor therapy have not recovered to CTCAE 5.0 Grade ≤ 1 before the administration (except for toxicity that is judged by the investigator to have no safety risk, such as alopecia, Grade 2 peripheral neurotoxicity and stable hypothyroidism with hormone replacement therapy).
13. Metastases to central nervous system or metastases to meninges.
14. History of other malignancy within 5 years of the enrollment (except for the following neoplastic diseases: adequately treated papillary thyroid carcinoma, cervix carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with radical surgery).
15. Active infection requiring systemic intravenous anti-infective therapy or fever of unknown origin exceeding 38℃ at enrollment.
16. Receiving therapeutic dosages of anticoagulants (except prophylactic anticoagulation) or history of bleeding ≥ Grade 3 within 3 months.
17. Subjects meet any of the following:

    * HIV infection (HIV antibody positive)
    * Active HBV infection (HBV DNA > 500 copies/mL or 100 IU/mL)
    * Active HCV infection (HCV antibody positive, HCV-RNA positive)
    * Treponema Pallidum infection (TP-Ab positive)
    * Subjects with known active tuberculosis (TB)
18. History of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    * Subjects with severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, II-III degree atrioventricular block.
    * According to New York Heart Association (NYHA) criteria, patients with grade II-IV cardiac insufficiency.
    * Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other Grade 3 or higher cardiovascular and cerebrovascular events within 6 months before the first dosage.
    * Clinically uncontrolled hypertension (systolic blood pressure > 140 mmHg and/or diastolic blood pressure > 90 mmHg despite optimal anti-hypertensive therapy).
    * Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, uncorrectable hypokalemia, congenital long QT syndrome, need to use any concomitant medication known to prolong the QT interval.
19. Clinically uncontrolled third space fluid
20. Known ≥ Grade 2 uveitis and retinopathy.
21. Subjects who are known to be allergic to IMB071703 injection or its excipients
22. Subjects with known, documented, or suspected drug abuse
23. Pregnant or lactating women
24. Subjects who, in the opinion of the investigator, have psychiatric disorders, poor compliance, inability to tolerate venous blood sampling, history of other serious systemic diseases, or other reasons that would make them inappropriate for participating in this clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Estimated)
Dates: Start 2023-02-24 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events/serious adverse event related with IMB071703 injection | From enrollment until 90 days after the last dose
Dose-limiting toxicity (DLT) | From the first dose of study drug up to 3 weeks
Maximum tolerated dose (MTD) and recommended phase II dose (RP2D) of IMB071703 injection | From first dose to disease progression or end of study, an average of 2 years

SECONDARY OUTCOMES:
Maximum measured plasma concentration (Cmax) of IMB071703 injection. | From first dose until 90 days after the last dose
Time to maximum plasma concentration (Tmax) of IMB071703 injection. | From first dose until 90 days after the last dose
Half-life (T1/2) of IMB071703 injection. | From first dose until 90 days after the last dose
Immunogenicity profile of IMB071703 injection. | From first dose until 90 days after the last dose
  Blood samples will be collected from subjects post treatment for assessment to detect the presence of anti-drug antibodies and neutralizing antibodies.
Objective Response Rate (ORR) | From first dose to disease progression or end of study, an average of 2 years
Duration of Response (DOR) | From first dose to disease progression or end of study, an average of 2 years
Disease control rate (DCR) | From first dose to disease progression or end of study, an average of 2 years
Progression free survival (PFS) | From first dose to disease progression or end of study, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oncology, Shanghai East Hospital, Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No